CLINICAL TRIAL: NCT02287584
Title: Confirmatory Study of DSP-5423P in Patients With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D4904020; JapicCTI-142688 (Registry Identifier: JAPIC Clinical Trials Informaton)
Record Dates: First submitted 2014-11-06; First posted 2014-11-10 (Estimated); Results first posted 2020-12-23 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- DSP-5423P Placebo (Placebo Comparator): Percutaneous DSP-5423P Placebo was applied once daily for 6 weeks during the double-blinded treatment phase. Subjects who completed the double-blind treatment phase were able to entere the open-label treatment phase. The study drug was applied to the back, chest, or abdomen.
  Interventions: Drug: DSP-5423P Placebo
- DSP-5423P 40mg (Experimental): Percutaneous DSP-5423P 40mg was applied once daily for 6 weeks during the double-blinded treatment phase. Subjects who completed the double-blind treatment phase were able to entere the open-label treatment phase. The study drug was applied to the back, chest, or abdomen.
  Interventions: Drug: DSP-5423P 40mg
- DSP-5423P 80mg (Experimental): Percutaneous DSP-5423P 80mg was applied once daily for 6 weeks during the double-blinded treatment phase. Subjects who completed the double-blind treatment phase were able to entere the open-label treatment phase. The study drug was applied to the back, chest, or abdomen.
  Interventions: Drug: DSP-5423P 80mg
- DSP-5423P Placebo-to-Flex (Experimental): Percutaneous Subjects received DSP-5423P Placebo once daily for 6 weeks in the double-blind treatment phase. In the open-label treatment phase, DSP-5423P was applied as flexible dose (40, 60, or 80 mg) once daily for 28 weeks (outside Japan) or 52 weeks (in Japan). The study drug was applied to the back, chest, or abdomen.
  Interventions: Drug: DSP-5423P Placebo-to-Flex
- DSP-5423P Active-to-Flex (Experimental): Percutaneous Subjects received DSP-5423P 40mg or 80mg once daily for 6 weeks in the double-blind treatment phase. In the open-label treatment phase, DSP-5423P was applied as flexible dose (40, 60, or 80 mg) once daily for 28 weeks (outside Japan) or 52 weeks (in Japan). The study drug was applied to the back, chest, or abdomen.
  Interventions: Drug: DSP-5423P Active-to-Flex

INTERVENTIONS:
Drug: DSP-5423P Placebo — DSP-5423P Placebo was applied to the subject's back, chest, or abdomen once daily
  Arms: DSP-5423P Placebo
Drug: DSP-5423P 40mg — DSP-5423P 40mg was applied to the subject's back, chest, or abdomen once daily
  Arms: DSP-5423P 40mg
Drug: DSP-5423P 80mg — DSP-5423P 80mg was applied to the subject's back, chest, or abdomen once daily
  Arms: DSP-5423P 80mg
Drug: DSP-5423P Placebo-to-Flex — DSP-5423P Placebo:
  DSP-5423P Placebo was applied to the subject's back, chest, or abdomen once daily
  DSP-5423P Flex:
  DSP-5423P 20mg, 60mg or 80mg was applied to the subject's back, chest, or abdomen once daily
  Arms: DSP-5423P Placebo-to-Flex
Drug: DSP-5423P Active-to-Flex — DSP-5423P Active:
  DSP-5423P 40mg or 80mg was applied to the subject's back, chest, or abdomen once daily
  DSP-5423P Flex:
  DSP-5423P 20mg, 60mg or 80mg was applied to the subject's back, chest, or abdomen once daily
  Arms: DSP-5423P Active-to-Flex

SUMMARY:
The primary objective of the study is to evaluate the efficacy of DSP-5423P compared with placebo in patients with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have schizophrenia diagnosed by DSM-5, diagnostic criteria
* Patients who are aged 18 years or older at informed consent
* Patient understands the objectives and procedures of the study and who provide written voluntarily consent to participate in the study, etc.

Exclusion Criteria:

* Patients who fall under a contraindication listed in the blonanserin (LONASEN) package insert
* Patients with Parkinson disease
* Patients who previously received blonanserin, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 580 (Actual)
Dates: Start 2014-12; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Director, Drug Development Division, Study Director — Sumitomo Pharma Co., Ltd.
Locations (8):
- 3 Sites, Beijing, Etc., China
- 53 Sites, Tokyo Etc., Japan
- 14 Sites, Kuala Lumpur, Etc., Malaysia
- 9 Sites, Manila, Etc., Philippines
- 8 Sites, Smolensk, Etc, Russia
- 7 Sites, Seoul, Etc., South Korea
- 6 Sites, Taipei, Etc., Taiwan
- 8 Sites, Poltava, Etc, Ukraine

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were conducted in 8 countries/region between December 2014 and October 2018.
Pre-assignment Details: In this study, 675 subjects provided informed consent, 580 of 606 subjects.
Groups:
- DSP-5423P Placebo-to-Flex: Percutaneous DSP-5423P Placebo was applied once daily for 6 weeks during the double-blinded treatment phase. Subjects who completed the double-blind treatment phase were able to entere the open-label treatment phase. The study drug was applied to the back, chest, or abdomen once daily.
  DSP-5423P 20 mg patches and DSP-5423P 40 mg patches were used in the open-label treatment phase. One or two patches of DSP-5423P was/were applied once daily to subjects for a further 28 weeks (outside Japan) or 52 weeks (in Japan). The initial dose of DSP-5423P in the open-label treatment phase was 40 mg/day. After DSP-5423P 40 mg/day application for about 1 week, DSP-5423P could be applied as flexible dose within a range from 40 mg/day to 80 mg/day.
- DSP-5423P 40mg-to-Flex: Percutaneous DSP-5423P 40mg was applied once daily for 6 weeks during the double-blinded treatment phase. Subjects who completed the double-blind treatment phase were able to entere the open-label treatment phase. The study drug was applied to the back, chest, or abdomen once daily.
  DSP-5423P 20 mg patches and DSP-5423P 40 mg patches were used in the open-label treatment phase. One or two patches of DSP-5423P was/were applied once daily to subjects for a further 28 weeks (outside Japan) or 52 weeks (in Japan). The initial dose of DSP-5423P in the open-label treatment phase was 40 mg/day. After DSP-5423P 40 mg/day application for about 1 week, DSP-5423P could be applied as flexible dose within a range from 40 mg/day to 80 mg/day.
- DSP-5423P 80mg-to-Flex: Percutaneous DSP-5423P 80mg was applied once daily for 6 weeks during the double-blinded treatment phase. Subjects who completed the double-blind treatment phase were able to entere the open-label treatment phase. The study drug was applied to the back, chest, or abdomen once daily.
  DSP-5423P 20 mg patches and DSP-5423P 40 mg patches were used in the open-label treatment phase. One or two patches of DSP-5423P was/were applied once daily to subjects for a further 28 weeks (outside Japan) or 52 weeks (in Japan). The initial dose of DSP-5423P in the open-label treatment phase was 40 mg/day. After DSP-5423P 40 mg/day application for about 1 week, DSP-5423P could be applied as flexible dose within a range from 40 mg/day to 80 mg/day.
Period: the Double-blind Phase
Arm/Group | DSP-5423P Placebo | DSP-5423P 40mg | DSP-5423P 80mg | DSP-5423P Placebo-to-Flex | DSP-5423P 40mg-to-Flex | DSP-5423P 80mg-to-Flex
Started (Subjects treated in the double-blind treatment phase) | 190 | 196 | 194 | 0 | 0 | 0
Completed | 138 | 149 | 161 | 0 | 0 | 0
Not Completed | 52 | 47 | 33 | 0 | 0 | 0
Not completed — Adverse Event | 17 | 17 | 12 | 0 | 0 | 0
Not completed — Lack of Efficacy | 18 | 8 | 8 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 17 | 17 | 11 | 0 | 0 | 0
Not completed — Pregnancy | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 3 | 0 | 0 | 0 | 0
Not completed — other reasons | 0 | 0 | 1 | 0 | 0 | 0
Period: the Open-label Phase
Arm/Group | DSP-5423P Placebo | DSP-5423P 40mg | DSP-5423P 80mg | DSP-5423P Placebo-to-Flex | DSP-5423P 40mg-to-Flex | DSP-5423P 80mg-to-Flex
Started (Subjects completed the double-blind treatment phase) | 0 | 0 | 0 | 138 | 149 | 161
Treated (Subjects treated in the open-label treatment phase) | 0 | 0 | 0 | 131 | 143 | 157
Completed | 0 | 0 | 0 | 81 | 87 | 104
Not Completed | 0 | 0 | 0 | 57 | 62 | 57
Not completed — Did not receive drug | 0 | 0 | 0 | 7 | 6 | 4
Not completed — Adverse Event | 0 | 0 | 0 | 15 | 12 | 16
Not completed — Lack of Efficacy | 0 | 0 | 0 | 8 | 3 | 7
Not completed — Lost to Follow-up | 0 | 0 | 0 | 4 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 18 | 29 | 21
Not completed — non-compliance | 0 | 0 | 0 | 2 | 5 | 1
Not completed — other reasons | 0 | 0 | 0 | 3 | 6 | 6

BASELINE CHARACTERISTICS:
Population: modified Intention-to-treat (mITT) population
Groups:
- Total: Total of all reporting groups
Arm/Group | DSP-5423P Placebo | DSP-5423P 40mg | DSP-5423P 80mg | Total
Number analyzed (Participants) | 189 | 196 | 192 | 577
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.5 (13.67) | 40.7 (13.34) | 40.7 (14.35) | 41.0 (13.77)
Age, Customized [Count of Participants; unit: Participants]
  <65 | 176 | 185 | 180 | 541
  >=65 | 13 | 11 | 12 | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 80 | 78 | 234
  Male | 113 | 116 | 114 | 343
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 189 | 196 | 192 | 577
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 161 | 167 | 165 | 493
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 28 | 29 | 27 | 84
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Korea | 7 | 7 | 7 | 21
  Japan | 51 | 55 | 56 | 162
  Philippines | 25 | 22 | 22 | 69
  China | 9 | 9 | 10 | 28
  Taiwan | 14 | 15 | 17 | 46
  Ukraine | 14 | 17 | 15 | 46
  Malaysia | 55 | 58 | 53 | 166
  Russia | 14 | 13 | 12 | 39
Positive and Negative Syndrome Scale (PANSS) total score [Mean (Standard Deviation); unit: units on a scale] — The PANSS is comprised of 30 items and 3 subscales: the Positive subscale assesses hallucinations, delusions, and related symptoms; the Negative subscale assesses emotional withdrawal, lack of motivation, and similar symptoms; and the General Psychopathology subscale addresses other symptoms such as anxiety, somatic concern, and disorientation. An anchored Likert scale from 1 to 7, where values of 2 and above indicate the presence of progressively more severe symptoms, is used to score each item. Individual items are then summed to determine scores for the 3 subscales, as well as a total score
  units on a scale | 99.5 (13.84) | 101.6 (15.55) | 101.5 (14.76) | 100.9 (14.75)

OUTCOME MEASURES:

1. Primary Outcome: Change in PANSS Total Score From Baseline at Week 6
Description: The Positive and Negative Syndrome Scale (PANSS) is an interview-based measure of the severity of psychopathology in adults with psychotic disorders. The measure is comprised of 30 items and 3 subscales: the Positive subscale assesses hallucinations, delusions, and related symptoms; the Negative subscale assesses emotional withdrawal, lack of motivation, and similar symptoms; and the General Psychopathology subscale addresses other symptoms such as anxiety, somatic concern, and disorientation. An anchored Likert scale from 1 - 7, where values of 2 and above indicate the presence of progressively more severe symptoms, is used to score each item. Individual items are then summed to determine scores for the 3 subscales, as well as a total score. The PANSS total score is the sum of all 30 items and ranges from 30 through 210. A higher score is associated with greater illness severity.
Time Frame: Week 6
Population: modified Intention-to-treat (mITT) population; Change in PANSS Total Score Using Mixed Model for Repeated Measures in the Double-Blind Treatment Phase
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | DSP-5423P Placebo | DSP-5423P 40mg | DSP-5423P 80mg
Number analyzed (Participants) | 189 | 196 | 192
units on a scale
  baseline mean(SD) | 99.5 (13.84) | 101.6 (15.55) | 101.5 (14.76)
  Change at Week 6 | -10.8 (1.47) | -16.4 (1.43) | -21.3 (1.41)
Statistical Analysis 1: Comparison: DSP-5423P Placebo vs DSP-5423P 40mg; Using Mixed Model for Repeated Measures; Test type: Superiority; p = 0.007, Mixed Models Analysis — adjusted p value, Hochberg procedure; Mean Difference (Final Values) = -5.6, 95% CI 2-sided [-9.6 to -1.6], Standard Error of Mean 2.04
Statistical Analysis 2: Comparison: DSP-5423P Placebo vs DSP-5423P 80mg; Test type: Superiority; p < 0.001, Mixed Models Analysis — adjusted p-value, Hochberg procedure; Mean Difference (Final Values) = -10.4, 95% CI 2-sided [-14.4 to -6.4], Standard Error of Mean 2.03

2. Secondary Outcome: Proportion of Subjects Who Achieve a Response, Defined as 20% or Greater Improvement From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score at Week 6
Description: The PANSS is an interview-based measure of the severity of psychopathology in adults with psychotic disorders. The measure is comprised of 30 items and 3 subscales: the Positive subscale assesses hallucinations, delusions, and related symptoms; the Negative subscale assesses emotional withdrawal, lack of motivation, and similar symptoms; and the General Psychopathology subscale addresses other symptoms such as anxiety, somatic concern, and disorientation. An anchored Likert scale from 1 7, where values of 2 and above indicate the presence of progressively more severe symptoms, is used to score each item. Individual items are then summed to determine a total score. The PANSS total score is the sum of all 30 items and ranges from 30 through 210. A higher score is associated with greater illness severity.
  The Last Observation Carried Forward (LOCF) endpoint is defined as the last data captured on Day 1 through 7 days after the final application of DSP-5423P.
Time Frame: Week 6 (LOCF)
Population: modified Intention-to-treat (mITT) population
Measure: Count of Participants; unit: Participants
Arm/Group | DSP-5423P Placebo | DSP-5423P 40mg | DSP-5423P 80mg
Number analyzed (Participants) | 189 | 196 | 192
Participants
  >=20% improvement from baseline | 80 | 99 | 107
  >=30% improvement from baseline | 52 | 72 | 80
  >=40% improvement from baseline | 32 | 49 | 55
  >=50% improvement from baseline | 15 | 25 | 40

3. Secondary Outcome: Treatment Continuation Rate at 28 Weeks and 52 Weeks
Description: Percentage of subjects who stay the study up to 28 weeks (196 days, all countries), and 52 weeks (364 days, in Japan) and its 95% confidence interval.
Time Frame: Open-Week 28 and Open-Week 52 in the open-label treatment phase
Population: Open-label population: all subjects who applied DSP-5423P at least once in the open-label treatment phase.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Groups:
- DSP-5423P 40 Mg-to-Flex: Percutaneous Subjects received DSP-5423P 40 mg once daily for 6 weeks in the double-blind treatment phase. In the open-label treatment phase, DSP-5423P was applied as flexible dose (40, 60, or 80 mg) once daily for 28 weeks (outside Japan) or 52 weeks (in Japan). The study drug was applied to the back, chest, or abdomen.
- DSP-5423P 80 Mg-to-Flex: Percutaneous Subjects received DSP-5423P 80 mg once daily for 6 weeks in the double-blind treatment phase. In the open-label treatment phase, DSP-5423P was applied as flexible dose (40, 60, or 80 mg) once daily for 28 weeks (outside Japan) or 52 weeks (in Japan). The study drug was applied to the back, chest, or abdomen.
Arm/Group | DSP-5423P Placebo-to-Flex | DSP-5423P 40 Mg-to-Flex | DSP-5423P 80 Mg-to-Flex
Number analyzed (Participants) | 131 | 143 | 157
percentage of subjects
  28 weeks (196 days, all countries) | 64.4 [55.7 to 72.2] | 62.9 [54.5 to 70.3] | 70.7 [62.9 to 77.2]
  52 weeks (364 days, in Japan): number analyzed (Participants) | 27 | 33 | 42
  52 weeks (364 days, in Japan) | 44.4 [23.4 to 63.6] | 51.5 [33.5 to 66.9] | 50.0 [34.2 to 63.9]

ADVERSE EVENTS:
Time Frame: Up to 58 weeks
Description: Safety population in the double-blind phase; The safety population consisted of all subjects who were randomized and applied the study drug at least once during the study.
  DSP-5423P dosed population in the open-label population; The DSP-5423P dosed population consisted of all subjects who applied DSP-5423P at least once during the study.
Groups:
- DSP-5423P Placebo-to-Flex: Percutaneous Subjects received DSP-5423P Placebo once daily for 6 weeks in the double-blind treatment phase. In the open-label treatment phase, DSP-5423P was applied as flexible dose (40, 60, or 80 mg) once daily for 28 weeks (outside Japan) or 52 weeks (in Japan). The study drug was applied to the back, chest, or abdomen.
  DSP-5423P Placebo-to-Flex: DSP-5423P Placebo:
  DSP-5423P Placebo was applied to the subject's back, chest, or abdomen once daily
  DSP-5423P Flex:
  DSP-5423P 20mg, 60mg or 80mg was applied to the subject's back, chest, or abdomen once daily
- DSP-5423P 40mg-to-Flex: Percutaneous Subjects received DSP-5423P 40mg once daily for 6 weeks in the double-blind treatment phase. In the open-label treatment phase, DSP-5423P was applied as flexible dose (40, 60, or 80 mg) once daily for 28 weeks (outside Japan) or 52 weeks (in Japan). The study drug was applied to the back, chest, or abdomen.
  DSP-5423P Active-to-Flex: DSP-5423P Active:
  DSP-5423P 40mg or 80mg was applied to the subject's back, chest, or abdomen once daily
  DSP-5423P Flex:
  DSP-5423P 20mg, 60mg or 80mg was applied to the subject's back, chest, or abdomen once daily
- DSP-5423P 80mg-to-Flex: Percutaneous Subjects received DSP-5423P 80mg once daily for 6 weeks in the double-blind treatment phase. In the open-label treatment phase, DSP-5423P was applied as flexible dose (40, 60, or 80 mg) once daily for 28 weeks (outside Japan) or 52 weeks (in Japan). The study drug was applied to the back, chest, or abdomen.
Arm/Group | DSP-5423P Placebo | DSP-5423P 40mg | DSP-5423P 80mg | DSP-5423P Placebo-to-Flex | DSP-5423P 40mg-to-Flex | DSP-5423P 80mg-to-Flex
All-Cause Mortality (participants affected / at risk) | 0/190 | 0/196 | 1/194 | 1/131 | 0/196 | 4/194
Serious Adverse Events (participants affected / at risk) | 9/190 | 8/196 | 10/194 | 18/131 | 24/196 | 29/194
Other Adverse Events (participants affected / at risk) | 45/190 | 62/196 | 76/194 | 60/131 | 108/196 | 111/194
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DSP-5423P Placebo (N=190) | DSP-5423P 40mg (N=196) | DSP-5423P 80mg (N=194) | DSP-5423P Placebo-to-Flex (N=131) | DSP-5423P 40mg-to-Flex (N=196) | DSP-5423P 80mg-to-Flex (N=194)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sudden death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bartholin's abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intervertebral discitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Comminuted fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Akathisia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Guillain-Barre syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abnormal behaviour (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aggression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catatonia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Psychiatric symptom (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 2 (2) | 1 (1) | 1 (1) | 4 (4) | 2 (2) | 1 (2)
Schizophrenia (Psychiatric disorders) | 4 (4) | 4 (4) | 2 (2) | 9 (9) | 10 (11) | 10 (11)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Choking (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Social stay hospitalisation (Social circumstances) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DSP-5423P Placebo (N=190) | DSP-5423P 40mg (N=196) | DSP-5423P 80mg (N=194) | DSP-5423P Placebo-to-Flex (N=131) | DSP-5423P 40mg-to-Flex (N=196) | DSP-5423P 80mg-to-Flex (N=194)
Constipation (Gastrointestinal disorders) | 5 (5) | 8 (9) | 8 (9) | 6 (8) | 8 (11) | 13 (18)
Salivary hypersecretion (Gastrointestinal disorders) | 1 (1) | 0 (0) | 4 (4) | 3 (3) | 5 (6) | 10 (12)
Application site erythema (General disorders) | 3 (4) | 11 (17) | 18 (33) | 8 (12) | 12 (22) | 23 (43)
Application site pruritus (General disorders) | 1 (1) | 10 (11) | 14 (14) | 4 (5) | 14 (15) | 19 (20)
Nasopharyngitis (Infections and infestations) | 8 (8) | 5 (8) | 9 (9) | 11 (11) | 14 (27) | 25 (32)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 4 (6) | 3 (3) | 7 (10) | 11 (14) | 5 (7)
Weight increased (Investigations) | 6 (6) | 3 (3) | 3 (3) | 16 (16) | 13 (13) | 13 (13)
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 7 (7) | 4 (4) | 5 (6) | 11 (12)
Akathisia (Nervous system disorders) | 2 (2) | 11 (11) | 19 (22) | 11 (14) | 22 (27) | 27 (34)
Bradykinesia (Nervous system disorders) | 0 (0) | 1 (1) | 6 (6) | 1 (1) | 6 (6) | 11 (11)
Headache (Nervous system disorders) | 5 (5) | 9 (10) | 7 (7) | 6 (6) | 13 (21) | 17 (35)
Tremor (Nervous system disorders) | 5 (5) | 8 (9) | 17 (18) | 9 (9) | 14 (15) | 27 (33)
Insomnia (Psychiatric disorders) | 9 (10) | 10 (12) | 10 (11) | 5 (28) | 22 (32) | 20 (29)
Schizophrenia (Psychiatric disorders) | 10 (10) | 6 (6) | 1 (1) | 3 (3) | 13 (13) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-05-08): https://cdn.clinicaltrials.gov/large-docs/84/NCT02287584/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-10): https://cdn.clinicaltrials.gov/large-docs/84/NCT02287584/SAP_001.pdf